CLINICAL TRIAL: NCT06172556
Title: The Role of Early Cerebral Edema and Hematoma Assessment in Aneurysmal Subarachnoid Hemorrhage (a-SAH) in Predicting Structural Brain Abnormalities in Cognitive Impairments
Brief Title: Early Brain Damage Assessment in Aneurysmal Subarachnoid Haemorrhage in Predicting Cognitive Impairment
Status: Completed | Type: Observational
Sponsor: Hebei Medical University (Other)
Responsible Party: Principal Investigator, Wang Mingdong, MD, Associate Professor， Associate Chief Physician, Hebei Medical University
Other Study IDs: ID: 2023-1001
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — brain CT& MRI
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endovascular coiling, Surgical clipping, Mix — Endovascular coiling, Surgical clipping, Mix

SUMMARY:
the goal of this type of study : observation study is to learn about cerebral edema and hematoma in aneurysmal subarachnoid hemorrhage the main questions it aims to answer are current clinical practices lack predictive models to identify early structural brain abnormalities affecting cognition.

DETAILED DESCRIPTION:
the development of a predictive model termed the a-SAH Early Brain Edema/Hematoma Compression Neural (Structural Brain) Networks Score System (SEBE-HCNNSS).

ELIGIBILITY:
Inclusion Criteria: first-ever stroke, diagnosed with SAH via CT scan within 24 - 48 hours or lumbar puncture; 2) age between 18 and 70 years; 3) Confirmation of cerebral aneurysm by digital subtraction angiography (DSA) and/or CT angiography (CTA); 4) absence of neurological or psychiatric disease history and each unruptured intracranial aneurysm patient must be admitted to the hospital in excellent preoperative and pre-interventional condition; 5) Informed consent is signed by the patient and/or family. 6)Clinical diagnosis of Alzheimer's Disease Must be able to swallow tablets.

-

Exclusion Criteria: 1) patients over 70 years old; 2) presence of neurological focal deficits or severe aphasia; 3) cognitive dysfunction or history of cognitive decline including craniotomy, antipsychotics, neurodegenerative diseases, and chronic subdural hematoma; 4) concurrent acute or chronic infections, corneal or pupillary abnormalities, severe autoimmune or systemic diseases such as rheumatic illnesses of the musculoskeletal system; 5) concurrent severe organic dysfunction; 6) patients with recurrent aneurysms or aneurysms not first diagnosed in our hospital; 7) diagnosis of major psychosis according to the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition criteria 8)Insulin dependent diabetes,9)Thyroid disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Han Chinese emergency call
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Description of subarachnoid blood on cranial CT | 24 - 48 hours
  No visible blood, no effacement, and no widening of the longitudinal fissure of the brain. Absence of visible sulci due to effacement, diffuse deposits, or thin layers of blood at specified brain locations (L-FPN or D-FPN or M-FPN or PN or ON or M-CIN or other), or widening of the longitudinal fissure. Localized/diffuse blood deposits (<1 mm thick) at specified locations (L-FPN or D-FPN or M-FPN or PN or ON or M-CIN or other) in each section, without visible sulci in those areas at two predetermined levels in each hemisphere. For specified locations (L-FPN or D-FPN or M-FPN or PN or ON or M-CIN or other) in each section, absence of visible sulci at two predetermined levels in each hemisphere or disruption of the grey-white matter junction, with blood pooling (<1 mm thick) in ventricles or cerebral pools (insular pools, circumferential pools, lateral fissure pools, interpeduncular pools, lateral ventricles). Disappearance of sulci at two predetermined levels in each hemisphere or local

CONTACTS AND LOCATIONS:
Overall Officials: Mingdong Wang, Principal Investigator — The First Hospital of Hebei Medical University
Locations (1):
- The First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

REFERENCES:
- [Derived] Wang MD, Fu QH, Ni A, Yuan YP, Li CH, Wang ZX, Wang H. The role of early cerebral edema and hematoma assessment in aneurysmal subarachnoid hemorrhage (a-SAH) in predicting early brain injury (EBI) and cognitive impairment: a case controlled study. Int J Surg. 2024 Jun 1;110(6):3166-3177. doi: 10.1097/JS9.0000000000001244. PMID 38445521